CLINICAL TRIAL: NCT03135106
Title: A Randomized, Open-Label, Parallel Group, Drug-drug Interaction Study to Evaluate the Effect of Fluconazole and Itraconazole on the Pharmacokinetics of Erdafitinib in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Fluconazole and Itraconazole on Erdafitinib Pharmacokinetics in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108299; 2017-000117-23 (EudraCT Number); 42756493EDI1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-04-14; First posted 2017-05-01 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — erdafitinib; Fluconazole; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A: Erdafitinib alone (Experimental): Participants will receive single 4 milligram (mg) oral dose of erdafitinib on Day 1 in a fasted state.
  Interventions: Drug: Erdafitinib
- Treatment B: Erdafitinib + Fluconazole (Experimental): Participants will receive 400 mg fluconazole once daily orally from Day 1 to Day 11 in a fasted state and on Day 5, a single 4-mg oral dose of erdafitinib will be administered 30+/-10 minutes after the intake of 400 mg fluconazole dose.
  Interventions: Drug: Erdafitinib; Drug: Fluconazole
- Treatment C: Erdafitinib + Itraconazole (Experimental): Participants will receive 200 mg itraconazole once daily orally from Day 1 to Day 11 and on Day 5, a single 4-mg oral dose of erdafitinib will be administered 30+/-10 minutes after the intake of 200 mg itraconazole dose.
  Interventions: Drug: Erdafitinib; Drug: Itraconazole

INTERVENTIONS:
Drug: Erdafitinib — A single 4-mg of erdafitinib tablet will be administered on Day 1 in Treatment A and on Day 5 in Treatment B and C.
  Other Names: G-024
Drug: Fluconazole — A 400-mg fluconazole orally (4*100 mg capsules) will be administered from Day 1 to Day 11.
  Arms: Treatment B: Erdafitinib + Fluconazole
Drug: Itraconazole — A 200-mg itraconazole orally (2*100 mg capsules) will be administered from Day 1 to Day 11.
  Arms: Treatment C: Erdafitinib + Itraconazole

SUMMARY:
The purpose of this study is to evaluate the effect of multiple doses of fluconazole (an inhibitor of cytochrome P450 [CYP] 2C9 and CYP3A) and itraconazole (an inhibitor of CYP3A4 and P-glycoprotein [P-gp]) on the pharmacokinetics of a single 4-milligram (mg) oral dose of erdafitinib in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy on the basis of physical examination, medical history, vital signs, and triplicate 12-lead electrocardiogram (ECG) performed at screening
* Be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, other specific tests, blood coagulation or hematology are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator. Healthy participants should be characterized by the following genotype regarding CYP2C9: *1/*1 (wild type), *1/*2 or *1/*3
* If a woman, must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening and on Day 1
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 3 months after the last study drug administration
* If a man who is sexually active, must agree to use a condom; and if a man who is sexually active with a woman of childbearing potential and who has not had a vasectomy, must agree to use a condom in combination with an adequate contraception method as deemed appropriate by the investigator, example, partner using effective contraception (defined as hormonal contraception [pill, patch, injection], intrauterine device, surgical sterilization) during the study and not to donate sperm for 5 months after the last study drug administration

Exclusion Criteria:

* History of or current clinically significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* History or current evidence of ophthalmic disorder, such as central serous retinopathy (CSR) or retinal vein occlusion, active wet age related macular degeneration, diabetic retinopathy with macular edema, uncontrolled glaucoma, corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation, or ulceration
* Clinically significant abnormal values for hematology or clinical chemistry at screening as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or triplicate 12-lead ECG at screening as deemed appropriate by the investigator
* Donated blood or blood products or had substantial loss of blood (more than 500 [milliliter]mL) within 3 months before the first study drug administration or intention to donate blood or blood products during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of Erdafitinib | Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 168, 336, 504 and 672 hours post-dose
  The Cmax is the maximum observed plasma analyte concentration.
Area Under the Plasma Analyte Concentration-time Curve From the Time of 0 to one Week Post-doses [(AUC)0-168h] of Erdafitinib | Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 168 hours post-dose
  Area under the plasma analyte concentration-time curve from time 0 to one week post-dose (168 hours).
Area Under the Plasma Analyte Concentration-time Curve From Time 0 to Time of the Last Observed Quantifiable Concentration [(AUC)0-last] of Erdafitinib | Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 168, 336, 504 and 672 hours post-dose
  [(AUC)0-last] is defined as area under the plasma analyte concentration-time curve from time 0 to time of the last observed quantifiable concentration (Clast).
Area Under the Analyte Concentration-Time Curve From Time 0 to Infinite Time [(AUC)0-infinity] of Erdafitinib | Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 168, 336, 504 and 672 hours post-dose
  [(AUC)0-infinity] is defined as the area under the analyte concentration-time curve from time 0 to infinite time, calculated as the sum of AUClast and Clast/lambda (z), in which Clast is the last observed quantifiable concentration and lambda (z) is the first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) as a Measure of Safety | From screening to end of study (approximately up to 61 days)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

REFERENCES:
- [Derived] Poggesi I, Li LY, Jiao J, Hellemans P, Rasschaert F, de Zwart L, Snoeys J, De Meulder M, Mamidi RNVS, Ouellet D. Effect of Fluconazole and Itraconazole on the Pharmacokinetics of Erdafitinib in Healthy Adults: A Randomized, Open-Label, Drug-Drug Interaction Study. Eur J Drug Metab Pharmacokinet. 2020 Feb;45(1):101-111. doi: 10.1007/s13318-019-00581-9. PMID 31673875